CLINICAL TRIAL: NCT00991367
Title: Efficacy of CICATRIX (Asian Gotu Kola or Pennywort) in the Treatment of Recent Post-surgical Scars
Brief Title: CICATRIX in the Treatment of Recent Post-surgical Scars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Alfredo Abreu Daniel PhD, "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0909-CU
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Post-surgical Scars
Keywords: Post-surgical scars; Asian Gotu Kola; Asian Pennywort
MeSH Terms: interventions — Cosmetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Cicatrix
  Interventions: Other: Cicatrix
- B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cicatrix — Dosage commensurate with surface to be treated. After washing and drying the affected area, a thin layer of CICATRIX (Topical use) will be applied on the lesion rubbing in different directions for 2 minutes, three times a day, for 4 weeks.
  Other Names: Cosmetic
  Arms: A
Other: Placebo — Dosage commensurate with surface to be treated. After washing and drying the affected area, a thin layer of PLACEBO (Topical use) will be applied on the lesion rubbing in different directions for 2 minutes, three times a day, for 4 weeks.
  Arms: B

SUMMARY:
The purpose of the study is to assess the efficacy of CICATRIX (Asian Gotu Kola or Pennywort) usage in the treatment of recent post-surgical scars. The duration of this double-blind placebo controlled phase 3 clinical trial will be 4 weeks. The estimated number of persons to be recruited and randomized for the study is 90.

ELIGIBILITY:
Inclusion Criteria:

* Recent (less than 48 hours) post-surgical wound

Exclusion Criteria:

* Post-surgical wound with sepsis
* Usage of steroids within 30 days
* Malignant neoplastic conditions
* Alcoholism
* Handicap and/or psychiatric condition preventing treatment accomplishment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Length of the post-surgical scar(s) measured by a millimetric ruler at week 4 (end of the treatment) | 4 weeks

SECONDARY OUTCOMES:
Occurrence of adverse effects at week 4 (end of the treatment) | 4 weeks
Photographs of lesions at week 4 (end of the treatment) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omara Lemus, MD, Principal Investigator — "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital
Locations (1):
- "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital, Havana, La Habana, Cuba